CLINICAL TRIAL: NCT03041064
Title: A Single Center, Randomized, Split Body and Split Face, Double-Blinded, Multiple Sun Exposure Evaluation of Sunscreens of SPF 50+ and Above Under Actual Use Conditions
Brief Title: Multiday Beach Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CO-1602 0409 2933-SACT
Record Dates: First submitted 2016-10-13; First posted 2017-02-02 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Erythema
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPF 50/SPF 100 (Experimental): SPF 50 assigned to left side of face and body. SPF 100 assigned to right side of face and body
  Interventions: Other: 50/100
- SPF 100/SPF 50 (Experimental): SPF 100 assigned to left side of face and body. SPF 50 assigned to right side of face and body
  Interventions: Other: 100/50

INTERVENTIONS:
Other: 50/100 — SPF
  Arms: SPF 50/SPF 100
Other: 100/50 — SPF
  Arms: SPF 100/SPF 50

SUMMARY:
This is a randomized, double-blinded, single-center, split body and split face, multiple natural sunlight exposure evaluation of two marketed sunscreens under actual use conditions in healthy volunteers. Eligible subjects will be randomized to two treatment randomization groups: Left SPF (Sun Protection Factor) 100+/Right SPF 50+ or Left SPF 50+/Right SPF 100+. Assessment of erythema and pigmentation will be performed at baseline and after all natural sunlight exposure periods which will occur on at the same beach location over the course of 5 consecutive days. Subjects will be suspended from further natural light exposure periods following the observation of sunburn at any exposed body site.

DETAILED DESCRIPTION:
Randomized, double-blinded, single-center, split body and split face, in use study under multiple exposures to natural sunlight conditions in healthy volunteers.

Each subject will be instructed to self-apply the test products to the designated exposure body/face sites as they normally would for sunburn protection while at the beach. Exposure sites will be limited through the duration of the study to the face, neck, arms including shoulders and legs from the top of the knee down. Each of the two products will be applied exclusively to the exposure sites on the designated side of the body for the duration of the study. Product labeling will include a color coded indicator of application side and a standard sunscreen drug facts label containing usage directions.

The difference in the level of sunburn (erythema) protection afforded and the level of UV (Ultraviolet) induced pigmentation (melanogenesis) response mediated by the typical usage of SPF 50+ and SPF 100+ sunscreens will be assessed by clinical evaluation. Erythema and melanogenic response will also be evaluated at fixed body site locations by diffuse reflectance spectroscopy (DRS) and chromameter assessment. Subject product usage will be tracked by recording tube weight before and after product use. Sunlight exposure behavior will be tracked by subject activity diaries.

Solar ultraviolet radiation conditions will be recorded on a centralized stationary radiometer.

Erythema protection afforded by the two products will be based on the bilateral sunburn comparison of matched exposure sites and the erythema score for each exposure area.

Success criteria will be demonstration of superior sunburn protection of SPF 100+ as compared to SPF 50+ as indicated by less sunburn on the SPF 100+ side than the SPF 50+ side (based on bilateral sunburn comparison).

Mediation of the UV induced pigmentation response afforded by the two products will be based on the bilateral pigmentation comparison of matched exposure sites and chromameter and DRS measurements.

All subjects will be evaluated at baseline and at the beginning of each day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-60 years old
* Phototypes I, II and III according to Fitzpatrick's classification
* Be willing to not apply any topical products (face/body) and cleanse (face/body) each morning prior to study visit.
* Be willing to use study test products in place of current sun protection topical skincare products (this includes make-up) during study hours.
* Be willing to have 1x1 cm sites marked on your skin. A total of 12 sites will be marked including four on the face. Face sites will be marked by the corners only.
* Be willing to refrain from using other sunscreen products, excessive sun exposure or tanning beds outside of the study visits.
* Be willing to refrain from using new face/body cleanser products and brands cannot be switched during the study.
* Be willing to refrain from using any new personal care products (e.g. makeup) or changing existing brands during the study.
* Be willing to not shave or use any hair removal method on your face/body within the 24 hours prior to first study visit and for the study duration.

Exclusion Criteria:

* Individuals with known allergies or sensitivities to sunscreens or common topical skincare products.
* Presence of sunburn (i.e. clinical erythema score greater than 0), suntan, scars, tattoos, active dermal lesions, dysplastic nevi, uneven skin tone, damaged/broken skin, or excessive body hair* on the areas of skin to be evaluated. The presence of nevi (other than dysplastic nevi), blemishes, or moles is acceptable if, in the investigator's judgment, they will not compromise the study and will not jeopardize the subject's safety. Beach umbrellas are not permitted. Sunglasses are acceptable.
* *Hair is permitted to cover the back of the neck but long hair should be pulled into a ponytail leaving ears uncovered for Visits 2-6.
* Presence of excessive pigmentation (pre-existing sun tan) or photodamage on the exposure sites to be evaluated.
* Notable bilateral pigmentation discrepancies between the matched left and right side exposure sites (e.g., left arm more pigmented that right arm).
* For study day mornings, Subject has applied, and refuses to remove prior to acclimation, any topical products (face/body) to the areas of skin to be evaluated.
* Individuals with CONTROLLED health conditions. These individuals may be included in the study at the discretion of the PI:
* Subjects with conditions that do not affect the skin, such as hypertension and hypercholesterolemia, could be enrolled when their health condition is managed through diet, medication, etc.
* Subjects with conditions, which might affect the skin, such as hyper/hypothyroidism, diabetes must be excluded, regardless whether their health condition is controlled or not.
* Subjects who are taking medication for chronic conditions (e.g., insulin, antihistamines, steroidal and non-steroidal anti-inflammatory drugs, antibiotics, etc...) - exception could be made for hypercholesterolemia as per point VI.
* Individuals with any disease or condition of the skin including photosensitivity disorders (e.g., active [i.e. flaring] eczema or psoriasis, skin cancer, polymorphic light eruption (PMLE), systemic lupus erythematous (SLE), xeroderma pigmentosa) that could interfere with the study or increase risk to the subject.
* Subjects who are taking medication for chronic conditions that may make a subject more sun sensitive (e.g., Tetracyclines, antifungals, certain diuretics, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Mean bilateral sunburn comparison over matched exposure sites and sun exposure periods | Days 1-7
  The clinical evaluator assessed exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure . Clinical evaluation assessed erythema via a side-by-side comparison of the three exposure areas (matched sites) utilizing the bilateral comparison score (L1 = Subject's Left side noticeably more sunburned than right side; 0 = No difference in sunburn; R1 = Subject's Right side noticeably more sunburned than left side
Mean erythema scores over exposure areas and exposure periods, calculated separately for the left and right sides of the body/face | Days 1-7
  Clinical evaluator independently assessed each side of each exposure area for erythema utilizing the erythema assessment score. Erythema score for each of the 6 exposure areas utilizing a scale of 0-4 with permission for intermediate (half-point) grades ( 0 = no burn; 1 = possible burn, not clearly defined; 2 = defined redness clearly caused by UV; 3 = severe sunburn with pronounced redness; 4 = edema and blisters).

SECONDARY OUTCOMES:
Clinical evaluation of bilateral sunburn (erythema) comparison by exposure site and exposure period. | Days 3-7
  The clinical evaluator assessed exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure . Clinical evaluation assessed erythema via a side-by-side comparison of the three exposure areas (matched sites) utilizing the bilateral comparison score (L1 = Subject's Left side noticeably more sunburned than right side; 0 = No difference in sunburn; R1 = Subject's Right side noticeably more sunburned than left side).
Mean clinically evaluated bilateral sunburn (erythema) comparison per subject by exposure period. | Days 3-7
  The clinical evaluator assessed subject for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure. Clinical evaluation assessed erythema via a side-by-side comparison of the three exposure areas (matched sites) utilizing the bilateral comparison score (L1 = Subject's Left side noticeably more sunburned than right side; 0 = No difference in sunburn; R1 = Subject's Right side noticeably more sunburned than left side).
Mean clinically evaluated bilateral sunburn (erythema) comparison over exposure period by matched exposure site. | Days 3-7
  The clinical evaluator assessed subject for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure. Clinical evaluation assessed erythema via a side-by-side comparison of the three exposure areas (matched sites) utilizing the bilateral comparison score (L1 = Subject's Left side noticeably more sunburned than right side; 0 = No difference in sunburn; R1 = Subject's Right side noticeably more sunburned than left side).
Clinically evaluated erythema score by exposure site and exposure period. | Days 3-7
  The clinical evaluator assessed each of the 6 exposure sites separately for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema. The erythema score was based on a 0-4 scale with permission for intermediate (half-point) grades (0=no burn, 1=Possible burn, not clearly defined, 2= Defined redness clearly caused by UV, 3= Severe sunburn with pronounced redness, 4= Edema and blisters).
Change from baseline in clinically evaluated erythema score by exposure site and exposure period. | Days 3-7
  The clinical evaluator assessed each of the 6 exposure sites separately for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure. The erythema score was based on a 0-4 scale with permission for intermediate (half-point) grades (0=no burn, 1=Possible burn, not clearly defined, 2= Defined redness clearly caused by UV, 3= Severe sunburn with pronounced redness, 4= Edema and blisters).
Mean clinically evaluated erythema score per subject by exposure period. | Days 3-7
  The clinical evaluator assessed each subject for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure. The erythema score was based on a 0-4 scale with permission for intermediate (half-point) grades (0=no burn, 1=Possible burn, not clearly defined, 2= Defined redness clearly caused by UV, 3= Severe sunburn with pronounced redness, 4= Edema and blisters).
Mean change from baseline in clinically evaluated erythema score per subject by exposure period. | Days 3-7
  The clinical evaluator assessed each subject for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure. The erythema score was based on a 0-4 scale with permission for intermediate (half-point) grades (0=no burn, 1=Possible burn, not clearly defined, 2= Defined redness clearly caused by UV, 3= Severe sunburn with pronounced redness, 4= Edema and blisters).
Mean clinically evaluated erythema score over exposure periods by matched exposure site | Days 3-7
  The clinical evaluator assessed each of the 6 matched exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure. The erythema score was based on a 0-4 scale with permission for intermediate (half-point) grades (0=no burn, 1=Possible burn, not clearly defined, 2= Defined redness clearly caused by UV, 3= Severe sunburn with pronounced redness, 4= Edema and blisters).
Mean change from baseline in clinically evaluated erythema score over exposure periods by matched exposure site. | Days 3-7
  The clinical evaluator assessed each of the 6 matched exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure. The erythema score was based on a 0-4 scale with permission for intermediate (half-point) grades (0=no burn, 1=Possible burn, not clearly defined, 2= Defined redness clearly caused by UV, 3= Severe sunburn with pronounced redness, 4= Edema and blisters).
Mean clinically evaluated bilateral pigmentation (melanogenesis) comparison by exposure site and exposure period. | Days 3-7
  The clinical evaluator assessed exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced erythema 12-24 hours after a period of sun exposure . Clinical evaluation assessed erythema via a side-by-side comparison of the three exposure areas (matched sites) utilizing the bilateral comparison score (L1 = Subject's Left side noticeably more sunburned than right side; 0 = No difference in sunburn; R1 = Subject's Right side noticeably more sunburned than left side).
Mean clinically evaluated bilateral pigmentation (melanogenesis) comparison over matched exposure sites and exposure period. | Days 3-7
  The clinical evaluator assessed each of the 3 matched exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation 12-24 hours after a period of sun exposure. Clinical evaluation assessed pigmentation by side-by-side comparison of each of the three exposed areas utilizing the bilateral comparison score (L1 = subject's left side noticeably more pigmented than right side; 0 = no difference in pigmentation; R1 = Subject's right side noticeably more pigmented than left side).
Mean bilateral pigmentation (melanogenesis) comparison per subject by exposure period. | Days 3-7
  The clinical evaluator assessed each subject for UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation 12-24 hours after a period of sun exposure Clinical evaluation assessed pigmentation by side-by-side comparison of each of the three exposed areas utilizing the bilateral comparison score (L1 = subject's left side noticeably more pigmented than right side; 0 = no difference in pigmentation; R1 = Subject's right side noticeably more pigmented than left side) for each subject.
Mean bilateral pigmentation (melanogenesis) comparison over exposure periods by matched exposure site. | Days 3-7
  The clinical evaluator assessed each of the 3 matched exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation 12-24 hours after a period of sun exposure. Clinical evaluation assessed pigmentation by side-by-side comparison of each of the three exposed areas utilizing the bilateral comparison score (L1 = subject's left side noticeably more pigmented than right side; 0 = no difference in pigmentation; R1 = Subject's right side noticeably more pigmented than left side).
Bilateral pigmentation (melanogenesis) comparison on Day 7 by matched exposure sites as well as per subject | Days 3-7
  The clinical evaluator assessed each of the 3 matched exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation 12-24 hours after a period of sun exposure . Clinical evaluation assessed pigmentation by side-by-side comparison of each of the three exposed areas utilizing the bilateral comparison score (L1 = subject's left side noticeably more pigmented than right side; 0 = no difference in pigmentation; R1 = Subject's right side noticeably more pigmented than left side) for each subject.
Mean chromameter measurements ∆L* ∆a* ∆b* scores by exposure site and over exposure period. | Days 3-7
  UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure was assessed via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site
Mean changes from baseline in chromameter measurements ∆L* ∆a* ∆b* scores by exposure site and over exposure period. | Days 3-7
  UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure was assessed via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site.
Mean chromameter measurement ∆L* ∆a* ∆b* scores over exposure sites and exposure periods. | Days 3-7
  UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure was assessed via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site.
Mean changes from baseline in chromameter measurement ∆L* ∆a* ∆b* scores over exposure sites and exposure periods | Days 3-7
  UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure was assessed via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site.
Mean chromameter measurements ∆L* ∆a* ∆b* per subject by exposure period | Days 3-7
  UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure was assessed via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site.
Mean changes from baseline in chromameter measurements ∆L* ∆a* ∆b* per subject by exposure period. | Days 3-7
  UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure was assessed via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site.
Mean chromameter measurements ∆L* ∆a* ∆b* over exposure period by site. | Days 3-7
  UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure was assessed via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site.
Mean change from baseline in chromameter measurements ∆L* ∆a* ∆b* over exposure period by site. | Days 3-7
  UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure was assessed via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site.
Chromameter measurements ∆L*, ∆a*, ∆b* scores at Day 7 by matched exposure site as well as per subject. This analysis will include all subjects irrespective of the number of exposure periods. | Days 3-7
  The clinical evaluator assessed matched exposure sites for UV (SPF 50+ and SPF 100+ sunscreen) induced pigmentation response 12-24 hours after a period of sun exposure via chromameter measurements providing quantitative readings (L*, a*, b* values) of the skin color at each designated measurement site.
Number of subjects suspended from subsequent sun light exposure due to sunburn, by exposure period and by sunscreen product that triggered the suspension. | Days 3-7
  Summary statistics will be presented along with a detailed data listing.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kohli I, Nicholson CL, Williams JD, Lyons AB, Seo I, Maitra P, Tian X, Atillasoy E, Lim HW, Hamzavi IH. Greater efficacy of SPF 100+ sunscreen compared with SPF 50+ in sunburn prevention during 5 consecutive days of sunlight exposure: A randomized, double-blind clinical trial. J Am Acad Dermatol. 2020 Apr;82(4):869-877. doi: 10.1016/j.jaad.2019.09.018. Epub 2019 Sep 19. PMID 31542406